CLINICAL TRIAL: NCT04202692
Title: Evaluation of the Performance and Safety of an Oral Formulation of Hyaluronic Acid With Chondroitin Sulphate and Magnesium Trisilicate (GERDOff® Plus) in Patients With Gastro-Esophageal Reflux Disease: A Double-blind, Placebo-controlled, Randomized, Cross-over Study
Brief Title: Effect of a Combination Oral Formulation of Hyaluronic Acid, Chondroitin Sulphate and Magnesium Trisilicate in Patients With Gastro-Esophageal Reflux Disease Not Fully Satisfied With Their Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PSC-DS MATRIX 19
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERDOff Plus (Experimental): Hyaluronic acid + chondroitin sulphate + magnesium trisilicate melt in mouth tablets (1100 mg). 1 tablet q.i.d. (three after meals, one before resting) for 3 consecutive weeks. After three weeks of wash-out period,patients will take either placebo or GERDOff Plus q.i.d. (three after meals, one before resting) for another three weeks.
  Interventions: Device: Hyaluronic acid with chondroitin sulphate and magnesium trisilicate, 1100 mg melt in mouth tablet; Device: Placebo 1100 mg, identically-looking melt in mouth tablet
- Placebo (Placebo Comparator): Placebo melt in mouth tablets (1100 mg). 1 tablet q.i.d. (three after meals, one before resting) for three consecutive weeks. After three weeks of wash-out period, patients will take either placebo or GERDOff Plus q.i.d. (three after meals, one before resting) for another three weeks.
  Interventions: Device: Hyaluronic acid with chondroitin sulphate and magnesium trisilicate, 1100 mg melt in mouth tablet; Device: Placebo 1100 mg, identically-looking melt in mouth tablet

INTERVENTIONS:
Device: Hyaluronic acid with chondroitin sulphate and magnesium trisilicate, 1100 mg melt in mouth tablet — 1 tablet q.i.d. (three after meals, one before resting) for 3 consecutive weeks
  Other Names: GERDOff Plus
Device: Placebo 1100 mg, identically-looking melt in mouth tablet — 1 tablet q.i.d. (three after meals, one before resting) for 3 consecutive weeks
  Other Names: GERDOff Plus placebo

SUMMARY:
This is a post-market, multi-center, double-blind, placebo-controlled, randomized, cross-over study with GERDOff Plus added on top of the current PPI treatment in patients with GERD. The aim of the study is to evaluate the performance of GERDOff Plus, a class III medical device, consisting in a hyaluronic acid, chondroitin sulphate and magnesium trisilicate, in addition to the PPIs, in patients with GERD not fully satisfied with their current treatment with PPIs.

Patients will receive either GERDOff Plus or placebo q.i.d. for 21 days followed by a wash-out period of 3 weeks. After the wash-out period, the patients will receive either placebo or GERDOff Plus respectively

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent (ICF): a written informed consent must be obtained prior to any study related procedure being performed
* Male and female out-patients aged 18 to 80 years
* GERD diagnosis confirmed through a validated questionnaire (GERDQ score ≥ 8).
* EGD endoscopy performed within 1 year before screening
* Patients in continuous or intermittent treatment with PPI for at least 1 year and continuously for at least 4 weeks prior to study entry
* Patients not fully satisfied with current PPI treatment (1-3 score on 5-points Likert scale)

Exclusion Criteria:

* Dyspeptic patients or patients with overlapping symptoms with GI diseases other than GERD
* Histological evidence of Barrett's oesophagus > 1 cm in EGD endoscopy
* Peptic stricture in EGD endoscopy
* Concurrent findings in the EGD endoscopy that might interfere with the participation to the study (e.g cancer, peptic ulcer) as judged by the investigator
* Known impaired kidney or liver function at screening
* Presence of any relevant severe condition or clinically relevant abnormal parameters that in the opinion of the investigator may interfere with the participation to the study
* Medication use (including H2 antagonists, alginates, baclofen, NSAIDS, prokinetics, antidepressants) that may interfere with GERD symptom assessment within 2 weeks before the start of the study or during the study
* Pregnancy or breast-feeding
* Females of childbearing potential not employing adequate contraceptive methods
* Active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment are also acceptable)
* History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent
* History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements
* Treatment with any investigational drug within the previous 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction | From baseline to the end of the respective 3-week treatment period
  The percentage of patients with an improvement of at least 2 points in the patient satisfaction measured with a 1 to 5 Likert scale (1 worst satisfaction, 5 best satisfaction)

SECONDARY OUTCOMES:
Change of weekly frequency of each symptom using the Gastro Esophageal Reflux Disease Questionnaire (GERDQ) questionnaire | From baseline to the end of the respective 3-week treatment period
  The reduction of weekly frequency score (points) for each symptom (score from 0 to 3, where higher scores mean a worse outcome) assessed by GERDQ questionnaire.
  Frequency score (points) for symptom: 0=0 day, 1=1 day, 2=2-3 days, 3=4-7 days;
  1. How often did you have a burning feeling behind your breastbone (heartburn)? 0 1 2 3
  2. How often did you have stomach contents (liquid or food) moving upwards to your throat or mouth (regurgitation)? 0 1 2 3
  3. How often did you have a pain in the centre of the upper stomach? 3 2 1 0
  4. How often did you have nausea? 3 2 1 0
  5. How often did you have difficulty getting a good night's sleep because of your heartburn and ⁄ or regurgitation? 0 1 2 3
  6. How often did you take additional medication for your heartburn and ⁄ or regurgitation, other than what the physician told you to take? (such as Tums, Rolaids, Maalox?) 0 1 2 3
Change of weekly global score of symptoms using the Gastro Esophageal Reflux Disease Questionnaire (GERDQ) questionnaire | From baseline to the end of the respective 3-week treatment period
  The reduction of global score of GERQ questionnaire (score from 0 to 18, where higher scores mean a worse outcome). Global score is obtained as sum score of the 6 items detailed in Outcome 2.
Change of the intensity of each symptom using the Reflux Symptom Index (RSI) questionnaire | From baseline to the end of the respective 3-week treatment period
  The reduction of score of each symptom (from 0 to 5, where 0 = No problem and 5 = Severe Problem) assessed by RSI questionnaire
  1. Hoarseness or a problem with voice
  2. Cleaning throat
  3. Excess throat mucus or postnasal drip
  4. Difficulty swallowing food, liquids, or pills
  5. Coughing after eating or after lying down
  6. Breathing difficulties or chocking episodes
  7. Troublesome or annoying cough
  8. Sensations of something sticking or a lump in the throat
  9. Heartburn, chest pain, indigestion or stomach acid coming up
Change of the global score using the Reflux Symptom Index (RSI) questionnaire | From baseline to the end of the respective 3-week treatment period
  The reduction of global score of RSI questionnaire (from 0 to 45, where higher scores mean a worse outcome). Global score is obtained as sum score of the 9 items detailed in Outcome 4.
Assessment of palatability | At the end of 3-week treatment period
  The score of taste through a 4-point qualitative scale (where 1 - taste as bad as possible, and 4 - taste as good as possible)
Evaluation of the intake of rescue medications | From V1 (randomization) to V4 (Day 63 +/- 2 days)
  The amount of rescue medications taken

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Diakonie Klinikum GmbH - Jung- Stilling Krankenhaus, Siegen, North Rhine-Westphalia
  - Klinikum Region Hannover (KRH) Klinikum Siloah, Hanover

IPD SHARING:
Plan to Share IPD: No